CLINICAL TRIAL: NCT06631326
Title: Hepatic Arterial Infusion Chemotherapy Plus Lenvatinib and PD-1 Inhibitors Versus Lenvatinib Plus PD-1 Inhibitors as First-line Treatment for High Tumor Burden Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: a Target Trial Emulation Study
Brief Title: HAIC in Combination With PD-1 Inhibitors and Lenvatinib for High Tumor Burden Advanced HCC (CHANCE2416)
Status: Completed | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Haibo Shao, Professor, MD, PhD, First Hospital of China Medical University
Other Study IDs: CHANCE2416
Record Dates: First submitted 2024-10-05; First posted 2024-10-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HCC - Hepatocellular Carcinoma; Hepatic Arterial Infusion Chemotherapy; BCLC Stage C Hepatocellular Carcinoma; Lenvatinib; PD-1 Inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HAIC plus Lenvatinib and PD-1 inhibitors: Each patient should receive at least 2 cycles of HAIC, 2 cycles of PD-1inhibitors and take at least 2 months of Lenvatinib. The interval between HAIC and Lenvatinib plus PD-1 inhibitors should be within 2 months.
  Interventions: Procedure: hepatic artery infusion chemotherapy; Drug: Lenvatinib + PD-1 monoclonal antibody
- Lenvatinib plus PD-1 inhibitors: Each patient should receive at least 2 cycles of PD-1 inhibitors and 2 months of Lenvatinib.
  Interventions: Drug: Lenvatinib + PD-1 monoclonal antibody

INTERVENTIONS:
Procedure: hepatic artery infusion chemotherapy — Hepatic arterial infusion chemotherapy including FOLFOX and RALOX
  Groups: HAIC plus Lenvatinib and PD-1 inhibitors
Drug: Lenvatinib + PD-1 monoclonal antibody — PD-1 inhibitors including Camrelizumab, Sintilimab, Tislelizumab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of hepatic arterial infusion chemotherapy (HAIC) in combination with PD-1 inhibitors and Lenvatinib in patients with high tumor burden advanced-stage hepatocellular carcinoma (HCC) with portal vein tumor thrombus (PVTT).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old;
2. Diagnosis of HCC was confirmed by histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Diseases (AASLD) guideline;
3. At least one measurable intrahepatic lesion as per the RECIST 1.1 criteria;
4. HCC staging of the patients are consistent with both the BCLC stage C and the CNLC stage IIIa.
5. Presence of PVTT;
6. Patients received a first-line lenvatinib+PD-1 (L+P) inhibitors combination or that of HAIC+lenvatinib+PD-1 inhibitors (H+L+P). More specifically, the administration of lenvatinib was concomitant with PD-1 inhibitors, and HAIC was performed either concurrently with, or up to 2 months before or after the L+P inhibitors combination therapy. Patients in the H+L+P group should undergo at least 2 cycles of HAIC, receive at least 2 cycles of PD-1 inhibiors and take at least 2 months of lenvatinib. Patients in the L+P group should receive at least 2 cycles of PD-1 inhibiors, and take at least 2 months of lenvatinib.
7. Child-Pugh class A or B7;
8. Tumor burden meets up to 7 out criteria.

Exclusion Criteria:

1. Patients who took anti-tumor treatments before the combination therapy;
2. With other malignant tumors;
3. incomplete data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high tumor burden advanced HCC with PVTT who received HAIC in combination with PD-1 inhibitors and Lenvatinib under real-world practice conditions.
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) (Overall) | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.
Progression free survival(PFS) of intra-hepatic lesions | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease of intra-hepatic lesions or death due to any cause, whichever occurs first.
Progression free survival(PFS) of extra-hepatic lesions | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented appearance of extra-hepatic lesions or death due to any cause, whichever occurs first.
Progression free survival(PFS) of portal vein tumor thrombus (PVTT) | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease of PVTT or death due to any cause, whichever occurs first.
Objective response rate(ORR) per RESCIST 1.1 | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
ORR per mRECIST | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR per mRECIST.
ORR of PVTT | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR of PVTT.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | Up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Shao, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The first hospital of China medical university, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu J, Zhang S, Shao H. Hepatic arterial infusion chemotherapy plus lenvatinib and PD-1 inhibitors versus lenvatinib plus PD-1 inhibitors as first-line treatment for hepatocellular carcinoma with high tumour burden and portal vein tumour thrombus (CHANCE 2416): study protocol of a multicentre, retrospective, target trial emulation design. BMJ Open. 2025 Sep 9;15(9):e099510. doi: 10.1136/bmjopen-2025-099510. PMID 40930561